CLINICAL TRIAL: NCT02685579
Title: The Effect of Obstructive Sleep Apnea Treatment on Dizziness, Vertigo
Acronym: OSATDV
Status: Withdrawn | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Oron Yahav, ENT Specialist, Wolfson Medical Center
Other Study IDs: 0103-15-WOMC
Record Dates: First submitted 2016-02-13; First posted 2016-02-18 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Sleep Apnea; Dizziness; Vertigo
MeSH Terms: conditions — Sleep Apnea Syndromes; Dizziness; Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Treatment of Obstructive Sleep Apnea-CPAP/BiPAP etc./Diet/surgery/life style changes

SUMMARY:
Obstructive Sleep Apnea may cause dizziness or vertigo through hypoxia of the vestibular nuclei in the brain. Treating sleep apnea may improve dizziness or vertigo.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Diagnosed with Sleep Apnea
* DHI score equals or over 16 points

Exclusion Criteria:

* Pregnant women
* Patients diagnosed with mental diseases
* Patients taking anti-vertigo medications
* Patients after CVA or with peripheral neuropathy
* Patients who suffered severe head trauma
* Patients with chronic renal failure
* Patients with malignancy at the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People coming to the Sleep Study Laboratory at the E. Wolfson Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory Score | 3 months
  A change in the DHI score after treatment (before treatment and after, 3 months in between)

SECONDARY OUTCOMES:
Romberg on foam test | 3 months
  A change in the time participants will stand without falling on a foam (before treatment and after, 3 months in between)

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Centre, Holon, Israel

IPD SHARING:
Plan to Share IPD: No